CLINICAL TRIAL: NCT03790332
Title: Phase 1/2 Dose Finding and Safety Study of Ibrutinib in Pediatric Subjects With Chronic Graft Versus Host Disease (cGVHD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1146-IM; 2017-004558-41 (EudraCT Number)
Record Dates: First submitted 2018-12-12; First posted 2018-12-31 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-05

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: cGVHD; chronic graft versus host disease; PCYC1146IM; Pediatric; GVHD; chronic; 1146; Pharmacyclics; PCYC; Imbruvica; Ibrutinib; Immunology; graft versus host disease; corticosteroids; prednisone; PCI32765; PCYC1146; refractory; new onset graft versus host disease; refractory graft versus host disease; moderate cGVHD; severe cGVHD; moderate chronic graft versus host disease; severe chronic graft versus host disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Graft vs Host Disease | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1/2 (Experimental): Part A: Subjects ≥1 to <12 years of age with moderate or severe cGVHD after failure of 1 or more lines of systemic therapy, will receive oral ibrutinib once daily to determine Recommended Pediatric Equivalent Dose (RPED).
  Part A Continuation: Subjects participating in Part A may continue receiving daily ibrutinib until the RPED is determined, at which time their dose may be adjusted to the RPED.
  Part B: Subjects ≥1 to <12 years of age( upper age limit is < 22 years) with moderate or severe cGVHD after failure of 1 or more lines of systemic therapy or with newly diagnosed moderate or severe cGVHD will be dosed at the RPED. Subjects ≥12 will be given 420mg orally ibrutinib once daily.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib capsule, tablet, or suspension administered orally once daily
  Other Names: IMBRUVICA®; PCI-32765

SUMMARY:
Dose Finding and Safety Study of Ibrutinib in Pediatric Subjects with Chronic Graft Versus Host Disease (cGVHD)

ELIGIBILITY:
Key Eligibility:

Inclusion Criteria:

1. Part A: Subjects with moderate or severe cGVHD after failure of 1 or more lines of systemic therapy
2. Part B: Subjects with moderate or severe cGVHD after failure of 1 or more lines of systemic therapy, or subjects with new onset moderate or severe cGVHD and in need of systemic immunosuppression
3. History of allogeneic stem cell transplantation
4. Age

   * Part A: ≥1 to <12 years of age at the time of enrollment
   * Part B: ≥1 to <22 years of age at the time of enrollment
5. Karnofsky or Lansky (subjects <16 years of age) performance status ≥60

Key Eligibility:

Exclusion Criteria:

1. Presence of single organ genito-urinary involvement as the only manifestation of cGVHD
2. Received an investigational agent within 28 days before enrollment.
3. Received donor lymphocyte infusion (DLI) within 56 days before enrollment
4. Progressive underlying malignant disease or active post-transplant lymphoproliferative disease
5. Any uncontrolled infection or active infection requiring ongoing systemic treatment
6. Known bleeding disorders
7. Active hepatitis C virus (HCV) or hepatitis B virus (HBV)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Part A- PK (measured by AUC) will be reported descriptively | Approximately 24 months
Part B- PK (measured by AUC) will be reported descriptively | Approximately 7 years
Number of patients with adverse events as a measure of safety and tolerability | Approximately 7 years

SECONDARY OUTCOMES:
Part A- Number of patients with adverse events as a measure of safety and tolerability | Approximately 24 months
Part A- Pharmacodynamic effects as measured by in vitro BTK occupancy will be reported descriptively | Approximately 24 months
Part A continuation cohort and Part B-Response rate at 24 weeks | Approximately 6 months after last subject in enrolled
Part A continuation cohort and Part B- Duration of response (DOR) | Up to 48 weeks
Part A continuation cohort and Part B-Overall survival (OS) | Approximately 5 years after last subject enrolled
Part A continuation cohort and Part B-Late Effects Surveillance | Up to 5 years post enrollment
Growth Parameter height in meters will be reported descriptively | Up to 5 years post enrollment
  Subjects will be monitored for growth and development
Growth Parameter weight in kilograms will be reported descriptively. | Up to 5 years post enrollment
  Subjects will be monitored for growth and development
Available immune reconstitution laboratory parameters will be reported descriptively | Up to 5 years post enrollment
  Subjects will be monitored for immune reconstitution
Late effects (Adverse events suspected to be related to treatment) will be quantified and reported descriptively | Up to 5 years post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Gauri Sunkersett, Study Director — Pharmacyclics LLC.
Locations (48):
- United States (20):
  - City of Hope, Duarte, California
  - Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, California
  - Children's Hospital, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Primary Children's Hospital, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Cancer Center for Children. The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - The Royal Children's Hospital, Parkville, Victoria
  - Sydney Children's Hospital, Randwick
- St. Anna Kinderspital, Vienna, Austria
- Canada (2):
  - children's and Women's Health Centre of British Columbia, Vancouver, British Columbia
  - CHU Sainte-Justine, Montreal, Quebec
- France (2):
  - CHU Nantes - Hopital Enfant Adolescent, Nantes
  - Hôpital Robert-Debré Ap-Hp, Paris
- Charite-Universitaetsmedizin Berlin, Berlin, Germany
- Israel (3):
  - Hadassah Medical Centre, Jerusalem
  - Schneider Children's Medical Center in Israel, Petah Tikva
  - The Edmond and Lily Safra Children's Hospital, Ramat Gan
- Italy (4):
  - U.O.C. Ematologia Oncoematologia Pediatrica, Pavia, PV
  - Fondazione MBBM-Clinica Pediatrica, Monza
  - Dipartimento di Onco-Ematologia e Terapia Cellulare e Genica, Roma
  - S.C. Farmacia Pediatrica - Presidio Ospedaliero Infantile Regina Margherita, Turin
- Princess Maxima Center, Utrecht, Netherlands
- Russia (2):
  - Federal State Budgetary Institution "Dmitry Rogachev National Medical Research Center of Pediatric Hematology, Oncology and Immunology, Moscow
  - Federal State Budgetary Educational Institution of Higher Professional Education "LP.Pavlov First Saint Petersburg State Medical, Saint Petersburg
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Saint Mary's Hospital, Seoul
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario Universitario La Paz, Madrid
- Safari Day Care, Great Ormond Street Hospital, London, Greater London, United Kingdom